CLINICAL TRIAL: NCT03662035
Title: Apatinib Combined With S-1 in the Second-line Treatment of Advanced Pancreatic Cancer
Acronym: ASPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Kequn Xu, Director, head of oncology department, principal investigator, clinical professor, Changzhou No.2 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChangzhouNo2
Record Dates: First submitted 2018-08-15; First posted 2018-09-07 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — apatinib; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm (Experimental): Apatinib and S-1 Patients will be offered with Apatinib (500mg/d) and S-1 (60mg/d for BSA<1.25m2, 80mg/d for 1.25<BSA<1.5m2, and 100mg for BSA >1.5m2) until their disease have progressed.
  Interventions: Drug: Apatinib; Drug: S-1

INTERVENTIONS:
Drug: Apatinib — Apatinib
  Patients with advanced pancreatic cancer after failure of first-line chemotherapy will receive Apatinib (500mg/d, orally) 30 minutes after meal with warm water.Take 21 days as a cycle, patients will receive this treatment until they have got disease progressed. Dose adjustment: with 3/4 level of adverse reactions, the dose should be lowered to 250 mg/d.
Drug: S-1 — S-1
  Patients will receive S-1 (60mg/d for BSA<1.25m2, 80mg/d for 1.25<BSA<1.5m2, and 100mg for BSA >1.5m2, orally) twice a day, once after breakfast and once after dinner, for 14 days, 7 days for suspension and 21 days as one cycle.

SUMMARY:
The aim of this study was to determine the efficacy and safety of apatinib combined with S-1 on advanced pancreatic cancer patients after failure of first-line chemotherapy.

DETAILED DESCRIPTION:
1. To observe the curative efficacy of apatinib and S-1 on patients by analyzing the data of overall survival (OS), complete remission (CR) or partial remission (PR), the rate of progression free survival (PFS), levels of CA19-9 and VEGFR in serum [Time Frame: Evaluation at 2 month intervals through study completion from the date of study entry until the date of progression, up to 1 year].
2. To observe any adverse events, including abnormal clinical symptoms and vital signs, abnormal laboratory examinations, and to record the clinical features, severity, occurrence time, duration, management and prognosis of all subjects during the clinical study, and to determine the correlation between these adverse events and the experimental drugs. . The safety of drugs used in advanced pancreatic cancer was evaluated by CTCAE v4.0

ELIGIBILITY:
Inclusion criteria:

* 18-70 years old;
* ECOG score: 0-2;
* Have confirmed metastatic or locally advanced unresectable pancreatic cancer;
* At least one measurable lesion according to the RECIST1.1 standard;
* First-line chemotherapy drugs do not include S-1 or fluorouracil drugs;
* Main organ functions meet the following standards:

  * Baseline blood routine (the inspection standard should meet the requirements of no blood transfusion and blood products within 14 days, no use of G-CSF and other hematopoietic stimulant correction) :

    * Hemoglobin>80g/L
    * The absolute neutrophil count (ANC) 1.5 x 109 / L;
    * Blood platelet (PLT)> 90 x 109 / L;
  * Baseline biochemical test shall meet the following standards:

    * T BIL < 1.5*ULN.
    * A LT and AST<2.5*ULN, and in patients with liver metastasis < 5*ULN;
    * Cr≤1.5*ULN.
    * Albumin is greater than or equal to 30g/L;
* Women of child-bearing age must already have access to reliable contraception. Pregnancy tests (serum or urine) were performed within 7 days prior to enrollment and the results were negative, and a reliable method of contraception was preferred 8 weeks after the trial period and the last drug administration;
* Subjects will voluntarily join the study and sign the informed consent.

Exclusion criteria:

* Clearly allergic to apatinib, S-1 or their excipients;
* There are various factors affecting oral drugs (including dysphagia, chronic diarrhea, intestinal obstruction, etc.);
* Serious heart diseases in the last six months, including :

  * angina;
  * myocardial infarction;
  * heart failure;
  * interphase of QTc >450ms;
  * any other heart diseases that were judged as unsuitable for the study;
* Combined with uncontrollable hypertension after drug treatment (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg);
* Complicated with other serious medical diseases, including cerebrovascular disease, uncontrolled infection, active peptic ulcer, intestinal obstruction, etc.;
* Metastasis of tumor central nervous system;
* Women during pregnancy and lactation;
* The patient has been diagnosed with other tumors in the past five years, except for the following situations: B. Cured basal cell carcinoma of the skin and cured orthotopic carcinoma of the cervix;
* The time from the last chemotherapy is shorter than 4 weeks or 5 half-life (the time taken is older), and the time from the last radiotherapy is shorter than 4 weeks;
* Use the experimental drug within 28 days before enrollment;
* Patients with grade 2 or above toxicity caused by the use of anti-tumor drugs before enrollment;
* Have mental disorders or a history of substance abuse;
* Other circumstances that the investigator deems inappropriate to participate in the study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | one year.
  Progression-free survival is defined as the time from registration to the earlier of death or disease progression.

SECONDARY OUTCOMES:
Overall Survival | one year.
  OS refers to the date of registration to the date of death for any cause.
Duration of response | one year.
  DOR refers to the time from the time the measurement first conforms to the CR or PR criteria (whichever is first measured) to the time the first true record of disease recurrence or progression (using the minimum measurements recorded in the trial as a reference for disease progression).
Objective response rate | one year.
  ORR refers to the proportion of patients whose tumors have shrunk to a certain extent for a certain period of time, including CR and PR cases
Disease Control Rate | one year.
  DCR refers to the percentage of patients with confirmed complete remission, partial remission, and disease stabilization (> 8 weeks) who can evaluate efficacy

IPD SHARING:
Plan to Share IPD: No